CLINICAL TRIAL: NCT00480935
Title: A Phase II, Single Arm, Prospective Study of Neoadjuvant Sutent for Patients With Renal Cell Carcinoma
Brief Title: A Study of Neoadjuvant Sutent for Patients With Renal Cell Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: poor recruitment
Sponsor: University Health Network, Toronto (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-0017-C
Record Dates: First submitted 2007-05-29; First posted 2007-05-31 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Renal Cell Carcinoma
Keywords: Localized; Renal Cell Carcinoma; Neoadjuvant; Sunitinib Malate (Sutent)
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sunitinib Malate (Sutent) (Experimental): Sutent will be given at 50 mg once daily for 4 consecutive weeks followed by a 2 week rest period to comprise a complete cycle of 6 weeks. Patients will then continue on Sutent for another cycle of 4 consecutive weeks
  Interventions: Drug: Sunitinib Malate (Sutent)

INTERVENTIONS:
Drug: Sunitinib Malate (Sutent) — Sutent will be given at 50 mg once daily for 4 consecutive weeks followed by a 1 week washout period. The dosage may change during the cycle due to possible drug toxicities. The nephrectomy will then take place following a one-week washout period.
  Other Names: Sutent

SUMMARY:
Study Hypothesis: Patients with local renal cell carcinoma who are treated neoadjuvantly with Sutent may show a radiologic response to the study drug (Sutent).

The study is looking at the neoadjuvant (pre-surgery) administration of Sutent in patients with localized kidney cancer. The purpose of this research is also to evaluate both the safety and effectiveness of Sutent in this patient population.

DETAILED DESCRIPTION:
Sutent will be given at 50 mg once daily for 4 consecutive weeks followed by a 1 week rest period. The dosage may change during the cycle due to possible drug toxicities. The nephrectomy will then take place following a one-week washout period. After surgery, patients will have follow-up visits at 6 weeks and 3 months. Patients will be followed for 3 years after completions to assess late toxicities, time to progression and progression-free survival.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed renal cell carcinoma with a component of clear (conventional) cell histology, which has been assessed with biopsy at screening.
* Locally confined tumour ≤ 7 cm
* Has not undergone nephrectomy and is a candidate for surgical treatment of renal cell carcinoma
* Male or female, 18 years of age or older
* ECOG performance status 0 or 1
* Adequate organ function as defined by the following criteria:

  * Serum aspartate transaminase (AST; serum glutamic oxaloacetic transaminase [SGOT]) and serum alanine transaminase (ALT; serum glutamic pyruvic transaminase [SGPT]) less than or equal to 2.5 x central laboratory upper limit of normal (CL-ULN), or AST and ALT less than or equal to 5 x CL ULN if liver function abnormalities are due to underlying malignancy
  * Total serum bilirubin less than or equal to 1.5 x CL-ULN
  * Absolute neutrophil count (ANC) greater than or equal to 1500/mL
  * Platelets greater than or equal to 100,000/mL
  * Hemoglobin greater than or equal to 9.0 g/dL
  * Serum calcium less than or equal to 12.0 mg/dL
  * Serum creatinine less than or equal to 1.5 x CL-ULN
  * Prothrombin time (PT) less than or equal to 1.5 x CL-ULN
* Signed and dated informed consent document indicating that the patient (or legally acceptable representative) has been informed of all pertinent aspects of the trial prior to enrollment
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures

Exclusion Criteria:

* Prior therapy of any kind for RCC (including nephrectomy, immunotherapy, chemotherapy, radiation, hormonal, or investigational therapy)
* Abnormal ECG- including long QT/QTc interval, AV block or arrythmia
* Tumour associated with local extension into adjacent tissues
* Tumour associated with renal/vena caval thrombus
* Tumour associated with lymphadenopathy (lymph node > 1 cm)
* Evidence of rapidly progressive disease or other factors requiring surgery to take place before the 12 weeks scheduled for neoadjuvant treatment
* Major surgery within 4 weeks of commencing study treatment
* Any toxicity with a NCI CTCAE grade 3 or 4
* Diagnosis of any second malignancy within the last 5 years, except for adequately treated basal cell carcinoma, squamous cell skin cancer, or in situ cervical cancer
* Evidence of metastatic renal cell carcinoma
* Any of the following within the 12 months prior to study drug administration: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, or pulmonary embolism
* Pre-existing thyroid abnormality with thyroid function that cannot be maintained in the normal range with medication
* Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness
* Current treatment on another clinical trial
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2007-10; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
To assess the radiologic response rate associated with 1 cycle of Sutent for neoadjuvant treatment of patients with renal cell carcinoma | 5 weeks

SECONDARY OUTCOMES:
To assess the change in tumour vascularity in response to 1 cycle of neoadjuvant treatment of patients with renal cell carcinoma | 5 weeks
To assess the change in expression of the following tissue markers; PDGF-alpha, PDGF-Beta, Flt-3, VEGFR and c-KIT, as compared to pre-treatment biopsy tissue as well as to stage, gender and age-matched controls | 5 weeks
To evaluate the safety and tolerability of Sutent given preoperatively | 5 weeks
To assess late toxicities, time to progression, progression free survival, and survival | 5 weeks - 3 years
A DNA microarray will be used for gene expression profiling of the tissue harvested at biopsy and surgery to investigate differential expression profiles and their association with Sutent sensitivity or resistance | 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Finelli, MD MSc FRCSC, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Princess Margaret Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Mickisch GH, Garin A, van Poppel H, de Prijck L, Sylvester R; European Organisation for Research and Treatment of Cancer (EORTC) Genitourinary Group. Radical nephrectomy plus interferon-alfa-based immunotherapy compared with interferon alfa alone in metastatic renal-cell carcinoma: a randomised trial. Lancet. 2001 Sep 22;358(9286):966-70. doi: 10.1016/s0140-6736(01)06103-7. PMID 11583750
- [Background] Motzer RJ, Rini BI, Bukowski RM, Curti BD, George DJ, Hudes GR, Redman BG, Margolin KA, Merchan JR, Wilding G, Ginsberg MS, Bacik J, Kim ST, Baum CM, Michaelson MD. Sunitinib in patients with metastatic renal cell carcinoma. JAMA. 2006 Jun 7;295(21):2516-24. doi: 10.1001/jama.295.21.2516. PMID 16757724
- [Background] Volpe A, Panzarella T, Rendon RA, Haider MA, Kondylis FI, Jewett MA. The natural history of incidentally detected small renal masses. Cancer. 2004 Feb 15;100(4):738-45. doi: 10.1002/cncr.20025. PMID 14770429
- [Background] Lamuraglia M, Escudier B, Chami L, Schwartz B, Leclere J, Roche A, Lassau N. To predict progression-free survival and overall survival in metastatic renal cancer treated with sorafenib: pilot study using dynamic contrast-enhanced Doppler ultrasound. Eur J Cancer. 2006 Oct;42(15):2472-9. doi: 10.1016/j.ejca.2006.04.023. Epub 2006 Sep 11. PMID 16965911
- [Background] Marzola P, Degrassi A, Calderan L, Farace P, Nicolato E, Crescimanno C, Sandri M, Giusti A, Pesenti E, Terron A, Sbarbati A, Osculati F. Early antiangiogenic activity of SU11248 evaluated in vivo by dynamic contrast-enhanced magnetic resonance imaging in an experimental model of colon carcinoma. Clin Cancer Res. 2005 Aug 15;11(16):5827-32. doi: 10.1158/1078-0432.CCR-04-2655. PMID 16115922